CLINICAL TRIAL: NCT06033105
Title: Vitamin D Deficiency As a Risk Factor for the Development and Malignant Transformation of Oral Lichen Planus: a Case-control Study
Brief Title: Vitamin D Deficiency As a Risk Factor for the Development and Malignant Transformation of Oral Lichen Planus
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Salsabeel A Afifi, PhD, Lecturer, Fayoum University
Other Study IDs: 2191982
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-09

CONDITIONS: Oral Lichen Planus; Vitamin D Deficiency
MeSH Terms: conditions — Lichen Planus, Oral; Vitamin D Deficiency | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 35 OLP patients
  Interventions: Device: ELISA
- Group B: 35 healthy controls.
  Interventions: Device: ELISA

INTERVENTIONS:
Device: ELISA — Enzyme-linked immunosorbent assay (ELISA) was used following manufacturer's instructions. This test uses a competitive ELISA-based technique that was designed to quantitatively determine the concentration of 1,25-dihydroxyvitamin D3/D2 in human serum.

SUMMARY:
To examine how a lack of vitamin D may increase the risk of developing oral lichen planus and its malignant progression while accounting for sex, food habits, sunlight, socioeconomic level, and psychological variables.

ELIGIBILITY:
Inclusion Criteria:

* (Group A) patients presenting with a clinical picture and histological findings that confirm the diagnosis of OLP
* (Group B) age, sex, and dietary habits matched healthy controls.

Exclusion Criteria:

* (1) subjects who have been receiving any kind of VD supplements, multivitamins, or any drug that may affect VD measurements
* (2) patients with suspected restoration-related or smokeless tobacco-related lesions.
* (3) patients with any systemic medical condition or pregnant females.
* (4) patients with VD toxicity (VD≥100 ng/ml).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting with a clinical picture and histological findings that confirm the diagnosis of OLP (Group A) and age, sex, and dietary habits matched healthy controls (Group B).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
serum vitamin D level in OLP | 1 month
  measured by ELISA

SECONDARY OUTCOMES:
serum vitamin D level in correlation with sex, dietary habits and sun exposure. | 1 month
  Questionnaire, measured in proportions
serum vitamin D level in correlation with socioeconomic status | 1 month
  Kuppuswamy's socioeconomic status scale
serum vitamin D level in correlation with Psychological factors | 1 month
  Depression Anxiety and Stress Scale 21 (DASS-21)

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Upon Request